CLINICAL TRIAL: NCT00891150
Title: Intravenous Oxytocin Use to Decrease Blood Loss During Cesarean Section. What is the Optimal Dose: A Randomized Blinded Trial
Brief Title: Oxytocin to Decrease Blood Loss During Cesarean Section
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: American University of Beirut Medical Center (Other)
Responsible Party: Principal Investigator, Dr. Labib Ghulmiyeh, Assistant Professor, American University of Beirut Medical Center
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: OGY.LB.01
Record Dates: First submitted 2009-04-30; First posted 2009-05-01 (Estimated); Last update posted 2013-03-06 (Estimated); Status verified 2013-03

CONDITIONS: Complications; Cesarean Section
MeSH Terms: interventions — Oxytocin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- oxytocin (Active Comparator): group 1 will receive oxytocin solutions with 20U/500ml during cesarean section
  Interventions: Drug: Oxytocin
- oxytocin2 (Active Comparator): group 2 will receive oxytocin solutions with 30U/500ml during cesarean section
  Interventions: Drug: Oxytocin
- oxytocin3 (Active Comparator): group 3 will receive oxytocin solutions with 40U/500ml during cesarean section
  Interventions: Drug: Oxytocin

INTERVENTIONS:
Drug: Oxytocin — Pre-mixed, oxytocin solutions with either 20U/500ml, 30U/500ml or 40U/500ml of Lactated Ringer's solution will be available in the pharmacy department. The bags will be identical in appearance. Each bag will be labeled with a study identification number, from which the pharmacy could determine the administered dose. Subjects as well as the medical providers will be blinded to the assignment of the solution used.
  Immediately after delivery of the infant, the study solution will be infused over 30 minutes using a continuous infusion pump (666 mU/min versus 999 mU/min versus 1332mU/min).
  Other Names: Pitocin

SUMMARY:
The goal of this study is to determine the best dose of a drug called oxytocin, that is usually used to stop bleeding during a delivery, when used during a cesarean delivery. It will be administered during cesarean section in order to decrease the amount blood loss. The investigators are proposing to have 3 groups of subjects each given a different safe dose of oxytocin and then to assess the effectiveness of each regimens on the amount blood lost during cesarean sections.This will let use know which is the best lowest dose needed.

DETAILED DESCRIPTION:
This trial will be a randomized, blinded controlled trial that will be conducted at the American University of Beirut Medical Center Labor and Delivery Unit.

Identification of candidates:

* All women admitted to the Delivery Suite for elective cesarean delivery or needing cesarean delivery for obstetric reasons will be invited to participate in the study.
* Women will then be approached by the research assistants and/or investigators who will explain the objectives of the study and will ask eligible women to participate in the trial and sign a consent form.

Study subjects will be randomized using a computer-generated random number sequence stratified by elective or emergency cesarean section. At surgery, a sealed opaque envelope containing the randomization number and data sheet will be opened for each consenting patient.

Interventions:

Pre-mixed, oxytocin solutions with either 20U/500ml, 30U/500ml or 40U/500ml of Lactated Ringer's solution will be available in the pharmacy department. The bags will be identical in appearance. Each bag will be labeled with a study identification number, from which the pharmacy could determine the administered dose. Subjects as well as the medical providers will be blinded to the assignment of the solution used.

Immediately after delivery of the infant, the study solution will be infused over 30 minutes using a continuous infusion pump (666 mU/min versus 999 mU/min versus 1332mU/min). The placenta will be delivered spontaneously with gentle cord traction. In the postanesthesia care unit, our practice is to give all patients a mixture of 30 U, 20 U and 10U of oxytocin to run consecutively in 1 L of lactated Ringer's solution at a rate of 125 mL/h (41.7 mU/min), which will be continued for a total of 24 hours.

Determination of the need for additional uterotonic agents will be made by the obstetrician and administered and recorded by the anesthesiologist. At the discretion of the surgical team, additional oxytocin could be added to the study solution (eg, 20 U) before requesting methylergonovine, 0.2 mg IM, or 15-methyl prostaglandin F2a 250 mg IM. Intramuscular methylergonovine maleate, and/or carboprost tromethamine will be available in the operating room and will be administered if needed. Ephedrine will be used to treat hypotension after delivery if the systolic blood pressure is >25 mm Hg below baseline.

We will be comparing the mean difference of preoperative hemoglobin vs. postoperative hemoglobin in each group. It will be referred to as delta Hemoglobin (Δ Hb).

In addition, we will be assessing several parameters including uterine tone, volume of blood lost and laparotomy pads number and weight among other data.

We will be performing multiple comparisons among the 3 groups specifically towards our primary outcome which is change or drop in hemoglobin from predelivery to postdelivery level.

The arm of the study with the lowest dose of pitocin and with the least amount of blood loss would probably be the optimal dose needed during a cesarean section for a patient that satisfies all the inclusion criteria of this trial.

In most institutions worldwide, a protocol is usually applied that states how much pitocin should be added to a 1 liter bag of NS or LR during cesarean section. It often ranges from 10 units to 40 units depending on the surgeons preference and uterine tone. The uterus is exteriorized most of the time during the surgery. The uterine tone does play a role in the choice of which dose id to be used(low versus high dose), however the optimal, most efficient dose with the least amount of side effects is yet to be determined. We are aiming to determine the optimal dose that will prevent the obstetricians from the additional use of other uterotonics (methergine, prostaglandins) that carries of by themselves unwanted side effects.

ELIGIBILITY:
Inclusion Criteria:

* Study subjects will be women delivering via an elective cesarean section at term
* All study subjects will have singleton gestation with no obstetric or medical complication.

Exclusion Criteria:

* Laboring women
* Multifetal gestation
* Prolonged oxytocin use (>12 hours)
* Hypertensive disorders
* Chorioamnionitis
* Suspected macrosomia
* Polyhydramnios
* History of postpartum Hemorrhage
* Clotting disorder
* Intake of magnesium sulfate
* Uterine fibroids
* Placenta previa
* Placental abruption
* Anticoagulation

Ages: 15 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 200 (Estimated)
Dates: Start 2012-07; Primary Completion 2013-02 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
The change in hemoglobin as a measure of blood loss. The change in hemoglobin is defined as the difference between the predelivery hemoglobin value and the postpartum value | 1 year

SECONDARY OUTCOMES:
The need for blood transfusion and the use of additional uterotonic agents, pad weight, pad count, estimated blood loss. | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Labib M Ghulmiyyah, MD, Principal Investigator — American University of Beirut Medical Center
Locations (1):
- American University of Beirut Medical Center, Beirut, Lebanon

REFERENCES:
- [Derived] Ghulmiyyah LM, Usta IM, Ghazeeri G, Taher N, Abu-Ghannam G, Tamim H, Nassar AH. Intravenous Oxytocin Use to Decrease Blood Loss during Scheduled Cesarean Delivery: A Randomized Double-Blinded Controlled Trial (OXYTRIAL). Am J Perinatol. 2017 Mar;34(4):379-387. doi: 10.1055/s-0036-1592130. Epub 2016 Sep 2. PMID 27588932